CLINICAL TRIAL: NCT00443131
Title: Adjuvant Justification Study of Candidate Malaria Vaccines (257049), Administered According to a 0, 1, 2 Months Schedule .
Brief Title: Characterisation of the Immune Responses of 2 Experimental Malaria Vaccines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 107731
Record Dates: First submitted 2007-03-02; First posted 2007-03-05 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Malaria
Keywords: Adjuvant; Malaria; Safety; Immunogenicity
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Group A (Experimental)
  Interventions: Biological: GSK Malaria vaccine 257049
- Group B (Experimental)
  Interventions: Biological: GSK Malaria vaccine 257049
- Group C (Experimental)
  Interventions: Biological: GSK Malaria vaccine 257049

INTERVENTIONS:
Biological: GSK Malaria vaccine 257049 — Three-dose vaccination by slow intramuscular injection. Three different formulations of this vaccine are tested (without adjuvant, with adjuvant AS01B, with adjuvant AS02A).

SUMMARY:
In this study, two experimental malaria vaccines (with adjuvants) are tested to evaluate and characterise how the vaccine exactly works on the immune system by comparing it to a control (without adjuvant). The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* A male or female between, and including, 18 and 45 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Have clinically normal laboratory values for creatinine, alanine aminotransferase (ALT), aspartate aminotransferase (AST), complete blood count (CBC) and differential at screening.
* Be seronegative for human immunodeficiency virus-1 and 2 (HIV 1/2) antibodies, HBsAg and hepatitis C virus (HCV) antibodies.
* Have anti HBs titre ≥ 10mIU/ml at screening.
* If the subject is female, she must be of non-childbearing potential or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the first vaccine dose.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within 30 days of the first dose of vaccine.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Any history of clinical malaria.
* Known exposure to malaria parasites within the previous 12 months.
* Planned travel to a malaria endemic region during the study period.
* History of allergic reactions or anaphylaxis to previous immunizations.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Personal history of autoimmune disease or subjects who describe a first-degree relative with clearly documented autoimmune disease.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine(s).
* Major congenital defects or serious chronic illness(es).
* Acute disease at the time of enrolment.
* History of any neurologic disorders or seizures.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Hepatomegaly, right upper quadrant abdominal pain or tenderness.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* History of previous exposure to experimental products containing any component of the vaccines used in this study.
* Pregnant or lactating female.
* History of chronic alcohol consumption and/or drug abuse.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-03-26; Primary Completion 2007-07-01 (Actual); Study Completion 2007-07-13 (Actual)

PRIMARY OUTCOMES:
Anti-CS antibody titers. | One month post Dose 3.

SECONDARY OUTCOMES:
Occurrence, intensity and relationship to vaccination of solicited local and general symptoms. | During the 7-day follow-up period following vaccination after each vaccine dose.
Occurrence, intensity and relationship to vaccination of unsolicited symptoms. | During the 30-day follow-up period following vaccination after each vaccine dose.
Occurrence of serious adverse events. | Up until 1 month post dose 3.
Antibody responses to the P. falciparum circumsporozoite (CS) antigen. | At Day 0, prior to dose 2, prior to dose 3 and 1 month post-dose 3.
Antibody responses to HBs antigen. | At Day 0, prior to dose 2, prior to dose 3 and 1 month post-dose 3
Frequency of CS and Hepatitis B surface agent (HBs)-specific CD4+ and CD8+ T cells expressing Th1 specific activation markers and cytokines. | At Day 0, prior to dose 2, prior to dose 3 and 1 month post-dose 3

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 107731 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107731 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 107731 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 107731 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 107731 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 107731 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register